CLINICAL TRIAL: NCT01082835
Title: Jiangzhuo Qinggan Prescription and Irbesartan in the Treatment of Essential Hypertension(Hepatogastric Damp-heat), Randomized, Parallel-controlled, Multi-center Clinical Study
Brief Title: Jiangzhuo Qinggan Prescription and Irbesartan in the Treatment of Essential Hypertension(Hepatogastric Damp-heat)Clinical Study
Acronym: JZQG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Guang'anmen Hospital, China Academy of Chinese Medical Sciences
Other Study IDs: 0081122
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Hypertension; Metabolic Syndrome
Keywords: Chinese herbs
MeSH Terms: conditions — Hypertension; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- the group of Jiangzhuo Qinggan prescription
- the group of irbesartan

SUMMARY:
Jangzhuo Qinggan prescription and irbesartan in the treatment of essential hypertension(Hepatogastric Damp-heat), randomized, parallel-controlled, multi-center clinical study.

DETAILED DESCRIPTION:
Charged by the five research centers in line with traditional Chinese medicine hepatogastric Damp-heat syndrome 240 cases have hypertension, and overweight, as well as blood lipid disorders or diabetes were randomly divided into Chinese herbal compound Jiangzhuo Qinggan prescription group and western medicine irbesartan group.The treatment groups were compared 4-week step-down and regulation of blood lipids, blood sugar effect.

ELIGIBILITY:
Inclusion Criteria:

1. Consistent with diagnosed hypertension, blood pressure, for 1-2 grade.
2. Aged 18-65 years old.
3. Body mass index (BMI) ≥ 24kg/m2, but <35 kg/m2.
4. Waist circumference ≥ 85cm (male) or waist circumference ≥ 80cm (women).
5. Comply with any of the following 3 : triglyceride (TG) elevated levels of:> 150mg/dl (1.7mmol / l), or has received appropriate treatment; high-density lipoprotein - cholesterol (HDL-C) levels reduced: Men <40mg/dl (0.9mmol / l), women <50mg/dl (1.1mmol / l), or has received appropriate treatment; fasting plasma glucose (FPG) increased: FPG ≥ 100mg/dl (5.6mmol / l ), or previously diagnosed type 2 diabetes or have received appropriate treatment.
6. Hepatogastric Damp-heat syndrome differentiation.
7. To sign informed consent.

Exclusion Criteria:

1. Has been used to control lipids, blood sugar drugs, but use the time for those below the 1 month.
2. Nearly 3 months, weight loss ≥ 5%.
3. Suffering from congenital heart disease, rheumatic heart disease, congestive heart failure, unstable angina, and had a myocardial infarction, percutaneous transluminal coronary angioplasty (PTCA) or off-line clinical significance of arrhythmia.
4. Bilateral renal artery stenosis, solitary kidney, serum creatinine> 133μmol / L .
5. Active liver disease, history of chronic persistent hepatitis, ALT> upper limit of normal.
6. Peptic ulcer or malabsorption syndrome .
7. With insulin-treated diabetes.
8. There is a history of appetite or abuse of laxatives by hyperthyroidism.
9. Pregnancy, pregnancy or breast-feeding women to prepare.
10. For those who are allergic Chinese medicine, allergic people.
11. Mentally ill.
12. Hyperkalemia in patients.
13. Cancer.
14. Occurred within the past 6 months who had a stroke or transient ischemic attack (TIA).
15. Nearly 3 months in patients receiving other clinical studies.
16. Alcohol and / or psychoactive substances, drug abuse and dependency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Combined metabolic syndrome in patients with essential hypertension
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-07 (Estimated); Study Completion 2010-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Medical University ,Dongzhimen Hospital, Beijing, Beijing Municipality
  - Beijing Medical University,Dongfang Hospital, Beijing, Beijing Municipality
  - China Academy of Chinese Medical Sciences,Guang'anmen Hospital, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences Fu Wai Cardiovascular Hospital, Beijing, Beijing Municipality
  - Capital University of Medical, Anzhen Hospital, Beijng, Beijing Municipality